CLINICAL TRIAL: NCT06021314
Title: Investigation of the Relationship Between Generalized Joint Hypermobility and Brace Efficiency in Adolescent Idiopathic Scoliosis
Brief Title: Brace Efficiency and Generalized Joint Hypermobility
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Collaborators: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Senay Cerezci Duygu, Asst. Prof., Saglik Bilimleri Universitesi
Other Study IDs: 2022-374
Record Dates: First submitted 2023-03-08; First posted 2023-09-01 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-08

CONDITIONS: Scoliosis Idiopathic; Hypermobility, Joint
MeSH Terms: conditions — Joint Instability | interventions — Braces

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adolescent Idiopathic Scoliosis
  Interventions: Other: Brace

INTERVENTIONS:
Other: Brace — Cheneau type scoliosis brace due to brace indication for adolecant idiopatic scoliosis

SUMMARY:
The goal of this observational study is to learn about effect of generalised joint hypermobility on the effectiveness of the brace in children with Adolesan Idiopatic Scoliosis and who use braces due to brace indication.

The main questions it aims to answer are:

* Does Generalized Joint Hypermobility have an effect on the amount of in-brace improvement achieved in children using braces?
* Does Generalized Joint Hypermobility have an effect on the change in the numerical variables related to scoliosis recorded in the out-brace measurement at the end of 6 months?

ELIGIBILITY:
Inclusion Criteria:

* Being under brace treatment due to the diagnosis of adolescent idiopathic scoliosis.
* Having a standing posterior-anterior radiograph before and during the brace use.
* Having a curve of 20 degree and above according to the Cobb angle.
* Confirmation of participation.

Exclusion Criteria:

• Having systemic diseases related to GJH (Ehlers-Danlos, Down, Marfan, Larsen).

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants who were diagnosed with adolescent idiopathic scoliosis and planned to use a cheneau type scoliosis brace.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Change of in-brace scoliosis angle | Measurement-1: Just before starting the brace use (Retrospectively)/ Measurement-2: In-brace condition at the 4th week of the brace use
  "Cobb angle" will be taken as reference to determine the scoliosis angle. For Cobb angle measurement, the angle between the upper border of the upper vertebra and the lower border of the lowest vertebra will be calculated.
  In order to determine change of scoliosis angle with brace use, the x-ray image taken just before starting to use the brace and the x-ray image taken while the brace is on the participant (in-brace condition) at the 4th week of brace usage will be evaluated. The difference between the two measurements will be recorded as change of in-brace scoliosis angle.
Generalised Joint Hypermobility | After participant being included in the study, latest at the 4th week of the brace use.
  A nine-degree "Beighton scale" will be used to determine the occurrence of generalized joint hypermobility. Additionally, a five-part questionnaire by Hakim and Graham will be used. Obtaining 4 or more points on Beighton scale and simultaneously at least 2 points in the ques-tionnaire by Hakim and Graham will be adopted as a criterion for generalized joint hypermobility diagnosis.

SECONDARY OUTCOMES:
Change of in-brace vertebral rotation | Measurement-1: Just before starting the brace use (Retrospectively)/ Measurement-2: In-brace condition at the 4th week of the brace use
  The evaluation of vertebral rotation on radiographs will be made using the Raimondi method regolo (Marrapese Editore-Demi S.r.1., Rome). In roimondi method; through the offset shadow, the widths of the vertebral body are measured in millimeters. The width of each vertebra is determined on the anterior-posterior X-ray at the most narrow spot, the so called vertebral waist. The convex-sided pedicle is marked and bisected longitudinally by a line. In order to determine the pedicle offset, the distance of this bisecting line to the convexsided waist of the vertebral body is evaluated. The value of vertebral rotation is obtained by inserting the width and the pedicle offset in the Raimondi method regolo. The difference between the two measurements will be recorded as in-brace improvement at scoliosis angle.
Change of in-brace spinal height | Measurement-1: Just before starting the brace use (Retrospectively)/ Measurement-2: In-brace condition at the 4th week of the brace use
  The distance between T1-S1 vertebral bodies in the x-ray image will be recorded in mm to determine the spinal height. The difference between the two measurements will be recorded as change of in-brace spinal height.
Change of in-brace global cronal balance | Measurement-1: Just before starting the brace use (Retrospectively)/ Measurement-2: In-brace condition at the 4th week of the brace use
  The distance between T the midpoint of the C7 vertebra and the central sacral vertical line (CSVL) in the x-ray image will be recorded in mm to determine the global cronal balance of spine. The difference between the two measurements will be recorded as change of in-brace global cronal balance.
Change of in-brace apical translation | Measurement-1: Just before starting the brace use (Retrospectively)/ Measurement-2: In-brace condition at the 4th week of the brace use
  The distance between the center of apical vertebra in the major curve and the sacral vertical line (CSVL) in the x-ray image will be recorded in mm to determine the global cronal balance of spine. The difference between the two measurements will be recorded as change of in-brace apical translation.
Brace compliance | in-brace condition at the 4th week of the brace use
  Daily usage hours and total brace usage time will be questioned retrospectively at the 4th week of brace use.

CONTACTS AND LOCATIONS:
Locations (1):
- Senay Cerezci Duygu, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cerezci-Duygu S, Yagci G, Nurdogan K, Demirkiran HG. Bracing Outcomes in Adolescent Idiopathic Scoliosis: The Role of Generalised Joint Hypermobility. J Paediatr Child Health. 2025 Sep;61(9):1423-1430. doi: 10.1111/jpc.70127. Epub 2025 Jun 26. PMID 40568822